CLINICAL TRIAL: NCT06338423
Title: Use of a Vacuum Mattress During Laparoscopic Sleeve Gastrectomy to Reduce the Concentration of Rhabdomyolysis Markers and Acute Renal Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Mateusz Wierdak, MD PD, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JagiellonianU-08
Record Dates: First submitted 2024-03-24; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Rhabdomyolysis; Acute Kidney Injury; Bariatric Surgery Candidate
MeSH Terms: conditions — Rhabdomyolysis; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vacuum Mattress Arm (Experimental): Patients will be operated in a beach chair position. The patient will ley on vacuum mattresses during the surgery.
  Patients' demographics, and perioperative data including age, gender, body mass index (BMI), smoking, ASA score, incidence of co-morbidities, compliance with ERABS protocol, amount of intraoperative blood loss, intraoperative complications, and surgery duration will be collected. Blood samples will be collected on first postoperative day to measure RML markers (myoglobin, creatine kinase, creatinine). Symptoms of RML, AKI and other complications were monitored for 30 days after surgery.
  Interventions: Device: vacuum mattress
- Standard Mattress arm (Other): Patients will be operated in a beach chair position. The patient will ley on standard mattresses during the surgery.
  Patients' demographics, and perioperative data including age, gender, body mass index (BMI), smoking, ASA score, incidence of co-morbidities, compliance with ERABS protocol, amount of intraoperative blood loss, intraoperative complications, and surgery duration will be collected. Blood samples will be collected on first postoperative day to measure RML markers (myoglobin, creatine kinase, creatinine). Symptoms of RML, AKI and other complications were monitored for 30 days after surgery.
  Interventions: Other: Standard Mattress

INTERVENTIONS:
Device: vacuum mattress — vacuum mattresses used to better positioning of the patient
  Arms: Vacuum Mattress Arm
Other: Standard Mattress — Standard Mattress
  Arms: Standard Mattress arm

SUMMARY:
This prospective clinical trial aimed to assess the usefulness of the usage of a vacuum mattress during laparoscopic sleeve gastrectomy (LSG) in the reduction of levels of rhabdomyolysis markers (myoglobin, creatine kinase, creatinine) and incidence of RML and AKI in the postoperative period.

Method Patients

A prospective clinical trial has been conducted between January 2015 and December 2022 in a tertiary referral University Hospital (Krakow, Poland). It is designed as a single-center, prospective trial with two intervention arms. During the study, we specified 3 periods:

* January 2015 - December 2016 - only standard mattresses were used
* January 2017 - December 2019 - both types of mattresses were used
* January 2020 - December 2022 - only vacuum mattresses were used

Participants Patients aged ≥18 were qualified for LSG due to obesity and divided The first group (Vacuum Mattress group) are those laid on vacuum mattresses during the surgery. The control group consisted of patients for whom a standard operating mattress was used during the surgery. Patients with preoperative chronic renal failure were excluded from the study. Other exclusion criteria were perioperative complications which required postoperative hospitalization at the Intensive Care Unit and Compliance with Enhanced Recovery After Bariatric Surgery (ERABS) Protocol < 85%.

Procedures and perioperative care All patients underwent LSG. Patients were operated in the beach chair position. In the study group, the patient was laid on vacuum mattresses during the surgery. In the case of control group patients, a standard operating mattress was used during the surgery. Perioperative care for all patients was in accordance with the ERABS protocol adopted in our center[]. Blood samples were collected on the first postoperative to measure RML markers (myoglobin, creatine kinase, creatinine). Symptoms of RML, AKI, and other complications were monitored for 30 days after surgery.

End Point Criteria The primary endpoint is the incidence of postoperative AKI or biochemical or clinical diagnosis of RML which required additional treatment.

Secondary endpoints is the concentrations of RML markers (myoglobin, creatine kinase, creatinine) on the first postoperative day

ELIGIBILITY:
Inclusion Criteria:

Patients aged ≥18 which will be qualified for LSG due to obesity

Exclusion Criteria:

Patients with preoperative chronic renal failure will be excluded from the study. Other exclusion criteria are perioperative complications which require postoperative hospitalization at the Intensive Care Unit and Compliance with Enhanced Recovery After Bariatric Surgery (ERAbSERABS ) Protocol < 85%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1184 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidance of Rhabdomyolisis(RML) And/OR Acute Kidnay Injury (AKI) | 30 day
  The primary endpoint is the incidence of postoperative AKI or biochemical or clinical diagnosis of RML which requireds additional treatment.

SECONDARY OUTCOMES:
Concentration of myoglobin marker | 1 day
Concentration of creatine kinase marker | 1 day
Concentration of creatinine marker | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University Mecical Collage, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No